CLINICAL TRIAL: NCT04704154
Title: A Multi-indication, Single-treatment Arm, Open-label Phase 2 Study of Regorafenib and Nivolumab in Combination in Patients With Recurrent or Metastatic Solid Tumors
Brief Title: A Trial to Learn Whether Regorafenib in Combination With Nivolumab Can Improve Tumor Responses and How Safe it is for Participants With Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Bristol Myers Squibb Co. and Ono Pharmaceutical Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21136; 2020-003359-13 (EudraCT Number)
Record Dates: First submitted 2021-01-08; First posted 2021-01-11 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumors
Keywords: Pancreatic Ductal Adenocarcinoma (PDAC); Head and Neck Squamous Cell Carcinoma (HNSCC); Esophageal Squamous Cell Carcinoma (ESCC); Glioblastoma Multiforme (GBM); Anaplastic Astrocytoma (AA); Biliary Tract Carcinoma (BTC); PD-1 inhibitor; nivolumab; regorafenib; multi-kinase inhibitor
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Esophageal Squamous Cell Carcinoma; Glioblastoma; Astrocytoma | interventions — regorafenib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Regorafenib+Nivolumab (Experimental): Parallel-cohort in adult participants with selected recurrent or metastatic tumors (HNSCC, ESCC, PDAC, BTC, and GBM/AA) who have been previously treated with one or more systemic therapy for the selected tumor indication.
  Interventions: Drug: Regorafenib, (Stivarga, BAY73-4506); Drug: Nivolumab (Opdivo)

INTERVENTIONS:
Drug: Regorafenib, (Stivarga, BAY73-4506) — Intake orally, starting with 3x 30 mg tablets every day (once daily.) for 21 days of every 28-day cycle (21 days on, 7 days off).
  If the starting dose is well tolerated dose can be escalated to 120 mg (4x30 mg tablets).
Drug: Nivolumab (Opdivo) — 480 mg administered on Day 1 of each treatment cycle.

SUMMARY:
Researchers are looking for a better way to treat people with solid tumors. Before a treatment can be approved for people to take, researchers do clinical trials to better understand its safety and how it works.

In this trial, the researchers want to learn about regorafenib taken together with nivolumab in a small number of participants with different types of tumors. These include tumors in the head and neck, the esophagus, the pancreas, the brain, and the biliary tract. The biliary tract includes gall bladder and bile ducts.

The trial will include about 200 participants who are at least 18 years old. All of the participants will take 90 mg of regorafenib as a tablet by mouth. The dose of regorafenib can be adjusted up to 120 mg or down to 60 mg by the doctor based on how well a participant tolerates treatment. All of the participants will receive 480 milligrams (mg) of nivolumab through a needle put into a vein (IV infusion).

The participants will take treatments in 4-week periods called cycles. They will take regorafenib once a day for 3 weeks, then stop for 1 week. In each cycle, the participants will receive nivolumab one time. These 4-week cycles will be repeated throughout the trial. The participants can take nivolumab and regorafenib until their cancer gets worse, until they have medical problems, or until they leave the trial. The longest nivolumab can be given is up to 2 years.

During the trial, the doctors will take pictures of the participants' tumors using CT or MRI and will take blood and urine samples. The doctors will also do physical examinations and check the participants' heart health using an electrocardiogram (ECG). They will ask questions about how the participants are feeling and if they have any medical problems.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed selected recurrent or metastatic solid tumor types that have progressed after treatment with standard therapies and for which there are no curative intent surgery or chemoradiation.
* Cohort 1: subjects with HNSCC (Head and neck squamous-cell carcinoma) who have not received prior PD-1/PD-L1 inhibitor therapy.
* Cohort 2: subjects with HNSCC who have progressed on or after prior systemic therapy, at least one of which included a PD-1/PD-L1 inhibitor alone or in combination with chemotherapy.
* Cohort 3: subjects with ESCC (Esophageal Squamous Cell Carcinoma) who progressed on or after platinum and/or fluoropyrimidine based regimen.
* Cohort 4: subjects with PDAC (Pancreatic ductal adenocarcinoma) who have progressed on or after gemcitabine or fluoropyrimidine based regimens.
* Cohort 5: subjects with BTC (Biliary tract carcinoma) (intrahepatic or extrahepatic cholangiocarcinoma or gall bladder cancer) who have progressed on gemcitabine or fluoropyrimidine or platinum therapy or a combination of these agents.
* Cohort 6: subjects with Grade IV GBM (Glioblastoma multiforme) or Grade III AA (Anaplastic astrocytoma) (World Health Organization [WHO] criteria) with unequivocal first progression after surgery followed by radiotherapy and temozolomide.
* Documented HPV (Human papilloma virus) / p16 status for oropharyngeal cancer.
* Capable of giving signed informed consent, including compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.
* Adult participants of legal maturity (18 years or older).
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 to 1.
* Adequate hematologic and organ function as assessed by the following laboratory tests performed within 7 d before start of study treatment including:

  * Total bilirubin ≤1.5 x the upper limit of normal (ULN). Total bilirubin (≤3 x ULN) is allowed if Gilbert's syndrome is documented
  * Alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤3 x ULN (≤5 x ULN for participants with liver involvement of their cancer)
* Measurable disease by baseline CT or MRI per RECIST 1.1 or RANO.
* Participants must consent to provide recent biopsy/tumor tissue of a primary tumor lesion or from metastases (e.g. liver, lung) for HNSCC (IO treated) for Stage 1 and 2 and in HNSCC (IO naïve) cohort for Stage 2.
* Anticipated life expectancy greater than 3 months.
* Be able to swallow and absorb oral tablets.

Exclusion Criteria:

* Presence of symptomatic central nervous system (CNS) metastases, leptomeningeal metastases or spinal cord compression. Previously-treated lesions should be stable for at least 6 weeks prior to study entry.
* Participants with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of start of study treatment.
* Prior therapy with PD-1/PD-L1 or cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) inhibitors, or any form of immunotherapy to treat cancer (except cohort 2).
* Cohort 2: More than one prior therapy with PD-1/PD-L1 or CTLA-4 inhibitors, or any other form of immunotherapy to treat cancer.
* ESCC:

  * patients with apparent tumor invasion on organs located adjacent to the esophageal disease (e.g., the aorta or respiratory tract).
  * patients who have previously received taxane agents for recurrent/metastatic cancer.
* GBM/AA

  * Primary tumors localized to the brainstem or spinal cord.
  * Presence of diffuse leptomeningeal disease or extracranial disease.
  * Participants requiring > 4 mg of dexamethasone or biologic equivalent per day to control symptoms related to brain tumor and cerebral edema within 21 days of starting study treatment.
* Participants who have known dMMR/MSI-H cancers or NTRK (tropomyosin receptor kinase) fusions.
* Prior therapy with regorafenib.
* Systemic anti-cancer treatment within 14 days or less than 5 half-lives (whichever is shorter) of the first dose of study treatment.
* Participants who have permanent discontinuation of PD-1/PD-L1 therapy due to toxicity.
* Arterial thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks) within 6 months before the start of study treatment. Active pulmonary emboli or deep vein thrombosis that are significant or not adequately controlled on anticoagulation regimen as per investigator's judgement.
* History of cardiac disorders as defined by:

  * Congestive heart failure ≥ New York Heart Association (NYHA) class 2:
  * Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months), myocardial infarction less than 6 months before start of study drug.
  * Uncontrolled cardiac arrhythmias.
* Poorly controlled hypertension, defined as a blood pressure consistently above 140/90 mmHg despite optimal medical management.
* Participants with an active, known or suspected autoimmune disease.
* History of (non-infectious) pneumonitis that required steroids, current pneumonitis or interstitial lung disease.
* Active infection > NCI-CTCAE Grade 2.
* Positive test (from historical data or tested during screening) for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Any positive test result for hepatitis B virus (HBV) or hepatitis C virus (HCV) indicating presence of virus, e.g. Hepatitis B surface antigen (HBsAg, Australia antigen) positive (except for participants on anti-viral therapy for HBV with a viral load < 100 IU/mL), or Hepatitis C antibody (anti-HCV) positive (except if HCV-ribonucleic acid [RNA] negative).
* Pregnancy or breast feeding.
* Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial or interfere with the participation for the full duration of the trial.
* Participants with a current or past history of interstitial lung disease or pulmonary fibrosis diagnosed based on imaging or clinical findings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2024-03-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (6):
  - City of Hope - Duarte Cancer Center, Duarte, California
  - Rocky Mountain Cancer Centers / Aurora, CO, Aurora, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Baylor Charles A. Sammons Cancer Center at Dallas, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Belgium (3):
  - Hôpital Erasme/Erasmus Ziekenhuis, Brussels
  - UZ Antwerpen, Edegem
  - CHU de Liège, Liège
- France (6):
  - Institut Bergonie - Unicancer Nouvelle Aquitaine, Bordeaux
  - UNICANCER - Centre Leon Berard (CLB), Lyon
  - APHP-Hopital la Pitie Salpetriere, Paris
  - Institut de Cancerologie Ouest - Saint-Herblain, Saint-Herblain
  - Institut Claudius Regaud - iUCT Oncopole, Toulouse
  - Gustave Roussy - Departement Oncologie-Radiotherapie, Villejuif
- Italy (5):
  - AUSL di Bologna_Istituto delle Scienze Neurologiche - UO Oncologia del Sistema Nervoso, Bologna, Emilia-Romagna
  - IRCCS Foundation Istituto Neurologico Carlo Besta, Milan, Lombardy
  - Humanitas Mirasole S.p.A. - Oncologia Medica ed Ematologia, Rozzano, Lombardy
  - Istituto Oncologico Veneto_Padova - UOC Oncologia 1, Padua, Veneto
  - ASST Grande Ospedale Metropolitano Niguarda - Oncologia Falck, Milan
- Japan (5):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Kobe University Hospital, Kobe, Hyōgo
  - Saitama Cancer Center, Kitaadachi-gun, Saitama
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
- South Korea (2):
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
- Taiwan (3):
  - Chi Mei Medical Center, Taikang, Tainan
  - China Medical University Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (4):
  - Royal Marsden NHS Trust (Surrey), Sutton, Surrey
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry, West Midlands
  - Beatson West of Scotland Cancer Centre, Glasgow
  - The Royal Marsden NHS Foundation Trust | The Royal Marden Hospital - The Royal Marsden Clinical Trials Unit (CTU), London

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/21136
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — https://www.clinicaltrialsregister.eu/ctr-search/search?query=21136

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 34 study centers in 8 countries/regions from 03 February 2021 (first patient first visit) to 29 March 2024 (last patient last visit)
Pre-assignment Details: 175 participants were enrolled and received study treatment. Participants were enrolled in 6 cohorts: HNSCC IO naïve (N=30), HNSCC IO treated (N=20), ESCC (N=30), PDAC (N=20), BTC (N=45), and GBM/AA (N=30)
Groups:
- HNSCC (IO Naive): Participants with confirmed recurrent or metastatic Head and Neck Squamous Cell Carcinoma (HNSCC) without Immune-oncology (IO), received 480 mg nivolumab intravenously on day 1 of every treatment cycle. Regorafenib was given as 30 mg tablets daily (QD) for 3 weeks of each treatment cycle (28 days cycle length) with a starting dose of 90 mg that could be escalated to 120 mg if well tolerated.
- HNSCC (IO Treated): Participants with confirmed recurrent or metastatic Head and Neck Squamous Cell Carcinoma (HNSCC) and with Immune-oncology (IO) treated, received 480 mg nivolumab intravenously on day 1 of every treatment cycle. Regorafenib was given as 30 mg tablets daily (QD) for 3 weeks of each treatment cycle (28 days cycle length) with a starting dose of 90 mg that could be escalated to 120 mg if well tolerated.
- ESCC: Participants with confirmed recurrent or metastatic Esophageal Squamous Cell Carcinoma (ESCC) received 480 mg nivolumab intravenously on day 1 of every treatment cycle. Regorafenib was given as 30 mg tablets daily (QD) for 3 weeks of each treatment cycle (28 days cycle length) with a starting dose of 90 mg that could be escalated to 120 mg if well tolerated.
- PDAC: Participants with confirmed recurrent or metastatic Pancreatic Duct Adenocarcinoma (PADC) received 480 mg nivolumab intravenously on day 1 of every treatment cycle. Regorafenib was given as 30 mg tablets daily (QD) for 3 weeks of each treatment cycle (28 days cycle length) with a starting dose of 90 mg that could be escalated to 120 mg if well tolerated.
- Biliary Tract Cancer (BTC): Participants with confirmed recurrent or metastatic BTC received 480 mg nivolumab intravenously on day 1 of every treatment cycle. Regorafenib was given as 30 mg tablets daily (QD) for 3 weeks of each treatment cycle (28 days cycle length) with a starting dose of 90 mg that could be escalated to 120 mg if well tolerated.
- GBM/AA: Participants with Glioblastoma Multiforme (GBM) or Anaplastic Astrocytoma (AA) received 480 mg nivolumab intravenously on day 1 of every treatment cycle. Regorafenib was given as 30 mg tablets daily (QD) for 3 weeks of each treatment cycle (28 days cycle length) with a starting dose of 90 mg that could be escalated to 120 mg if well tolerated.
Period: Overall Study
Arm/Group | HNSCC (IO Naive) | HNSCC (IO Treated) | ESCC | PDAC | Biliary Tract Cancer (BTC) | GBM/AA
Started (Assigned to treatment) | 30 | 20 | 30 | 20 | 45 | 30
Completed (Ongoing with treatment till primary completion cut-off) | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 30 | 20 | 30 | 20 | 45 | 30
Not completed — Adverse Event | 3 | 2 | 4 | 2 | 3 | 0
Not completed — Death | 3 | 0 | 0 | 0 | 3 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 0 | 2 | 0
Not completed — Participant Decision | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 19 | 17 | 20 | 18 | 36 | 30
Not completed — Completed max. allowed treatment. A max. of 24 infusions of Nivolumab were allowed for participants | 2 | 0 | 1 | 0 | 1 | 0
Not completed — Patient continued in rollover study for regorafenib | 1 | 0 | 4 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): all participants who received study treatment were included in the full analysis set
Groups:
- HNSCC (IO Naive): Participants with confirmed recurrent or metastatic HNSCC and IO naive, received regorafenib in combination with nivolumab. (treatment details refers to Description under Participant Flow section above)
- HNSCC (IO Treated): Participants with confirmed recurrent or metastatic HNSCC and with IO treated, received regorafenib in combination with nivolumab. (treatment details refers to Description under Participant Flow section above)
- ESCC: Participants with confirmed recurrent or metastatic ESCC received regorafenib in combination with nivolumab. (treatment details refers to Description under Participant Flow section above)
- PDAC: Participants with confirmed recurrent or metastatic PADC received regorafenib in combination with nivolumab. (treatment details refers to Description under Participant Flow section above)
- Biliary Tract Cancer (BTC): Participants with confirmed recurrent or metastatic BTC received regorafenib in combination with nivolumab. (treatment details refers to Description under Participant Flow section above)
- GBM/AA: Participants with GBM or AA received regorafenib in combination with nivolumab. (treatment details refers to Description under Participant Flow section above)
- Total: Total of all reporting groups
Arm/Group | HNSCC (IO Naive) | HNSCC (IO Treated) | ESCC | PDAC | Biliary Tract Cancer (BTC) | GBM/AA | Total
Number analyzed (Participants) | 30 | 20 | 30 | 20 | 45 | 30 | 175
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 16 | 10 | 17 | 13 | 17 | 22 | 95
  65-<75 years | 12 | 4 | 11 | 7 | 22 | 7 | 63
  75-<85 years | 2 | 6 | 2 | 0 | 6 | 1 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 3 | 11 | 20 | 10 | 55
  Male | 25 | 14 | 27 | 9 | 25 | 20 | 120
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 15 | 11 | 21 | 5 | 11 | 2 | 65
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 6 | 6 | 7 | 13 | 27 | 26 | 85
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 9 | 3 | 2 | 2 | 6 | 2 | 24

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Tumor response was evaluated as ORR per RECIST 1.1 by local assessments for all tumor types, except for GBM/AA, where ORR per RANO by local assessment was used. ORR was defined as the proportion of participants with best overall response of complete response (CR) or partial response (PR). Participants for whom best overall tumor response was not CR or PR, as well as participants without any post-baseline tumor assessment were considered non-responders. Descriptive statistics were done, no inferential statistical analyses were performed.
Time Frame: From first participant enrolled to cut-off date (ie after the last participant has been followed for approximately 10 months) approximately 26 months
Population: FAS: all participants who received study treatment were included in the full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | HNSCC (IO Naive) | HNSCC (IO Treated) | ESCC | PDAC | Biliary Tract Cancer (BTC) | GBM/AA
Number analyzed (Participants) | 30 | 20 | 30 | 20 | 45 | 30
Participants | 6 | 1 | 15 | 0 | 2 | 1

2. Secondary Outcome: Duration of Response (DOR)
Description: Defined as the time (in days) from the first documented objective response of PR or CR, whichever is noted earlier, to disease progression or death (if death occurs before progression is documented). DOR will be defined for responders only, i.e. participants with a CR or PR.
Time Frame: as for outcome 1
Population: Subgroup of participants that had a best overall response of CR or PR that had received the study treatment
Measure: Median (80% Confidence Interval); unit: Days
Arm/Group | HNSCC (IO Naive) | HNSCC (IO Treated) | ESCC | PDAC | Biliary Tract Cancer (BTC) | GBM/AA
Number analyzed (Participants) | 6 | 1 | 15 | 0 | 2 | 1
Days | NA [654 to NA] — Value cannot be estimated due to censored data, insufficient number of participants with events | NA [NA to NA] — Value cannot be estimated due to censored data, insufficient number of participants with events | 420 [112 to 617] |  | 432 [112 to NA] — Value cannot be estimated due to censored data, insufficient number of participants with events | 140 [NA to NA] — Value cannot be estimated due to censored data, insufficient number of participants with events

3. Secondary Outcome: Disease Control Rate (DCR)
Description: CR = Complete response; PR = Partial response; SD = Stable disease
Time Frame: as for outcome 1
Population: FAS: all participants who received study treatment were included in the full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | HNSCC (IO Naive) | HNSCC (IO Treated) | ESCC | PDAC | Biliary Tract Cancer (BTC) | GBM/AA
Number analyzed (Participants) | 30 | 20 | 30 | 20 | 45 | 30
Participants | 16 | 13 | 22 | 7 | 24 | 10

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time (in days) from the start of study intervention to the date of first objectively documented progressive disease (PD) or death from any cause (if no progression was documented).
Time Frame: as for outcome 1
Population: FAS: all participants who received study treatment were included in the full analysis set
Measure: Median (80% Confidence Interval); unit: Days
Arm/Group | HNSCC (IO Naive) | HNSCC (IO Treated) | ESCC | PDAC | Biliary Tract Cancer (BTC) | GBM/AA
Number analyzed (Participants) | 30 | 20 | 30 | 20 | 45 | 30
Days | 79 [50 to 227] | 105 [52 to 115] | 259 [110 to 472] | 53 [48 to 111] | 98 [55 to 112] | 55 [52 to 84]

5. Secondary Outcome: 6 Months PFS
Description: 6 Months PFS rate
Time Frame: Up to last participant follow 6 months (approximately 22 months)
Population: FAS: all participants who received study treatment were included in the full analysis set
Measure: Number (80% Confidence Interval); unit: Proportion of participants
Arm/Group | HNSCC (IO Naive) | HNSCC (IO Treated) | ESCC | PDAC | Biliary Tract Cancer (BTC) | GBM/AA
Number analyzed (Participants) | 30 | 20 | 30 | 20 | 45 | 30
Proportion of participants | 0.455 [0.337 to 0.573] | 0.263 [0.134 to 0.393] | 0.533 [0.417 to 0.650] | 0.050 [0.000 to 0.112] | 0.148 [0.077 to 0.218] | 0.167 [0.079 to 0.254]

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time (in days) from the start of study intervention to the date of death due to any cause.
Time Frame: as for outcome 1
Population: FAS: all participants who received study treatment were included in the full analysis set
Measure: Median (80% Confidence Interval); unit: Days
Arm/Group | HNSCC (IO Naive) | HNSCC (IO Treated) | ESCC | PDAC | Biliary Tract Cancer (BTC) | GBM/AA
Number analyzed (Participants) | 30 | 20 | 30 | 20 | 45 | 30
Days | 358 [198 to 418] | 355 [126 to 614] | 627 [431 to 865] | 259 [134 to 311] | 246 [176 to 386] | 245 [127 to 377]

7. Secondary Outcome: 1 Year OS
Time Frame: From first participant enrolled to cut-off date (ie after the last participant has been followed for approximately 10 months) approximately 26 month]
Population: FAS: all participants who received study treatment were included in the full analysis set
Measure: Number (80% Confidence Interval); unit: Proportion of participants
Arm/Group | HNSCC (IO Naive) | HNSCC (IO Treated) | ESCC | PDAC | Biliary Tract Cancer (BTC) | GBM/AA
Number analyzed (Participants) | 30 | 20 | 30 | 20 | 45 | 30
Proportion of participants | 0.415 [0.298 to 0.532] | 0.444 [0.294 to 0.595] | 0.764 [0.664 to 0.864] | 0.281 [0.145 to 0.418] | 0.422 [0.323 to 0.521] | 0.337 [0.223 to 0.451]

8. Secondary Outcome: Number of Participants With Adverse Events
Description: AEs were considered to be treatment-emergent (TEAEs) if they started or worsened after the start of first study drug administration until 30 days after regorafenib treatment discontinuation or 100 days after the last dose of nivolumab, whatever occurred later.
Time Frame: Up to the last participant has been followed for approximately 10 months, summed up to approximately 26 months
Population: Safety analysis set (SAF): all participants who received study treatment were included in the safety analysis set. As the safety analysis set equals the full analysis, all safety related analysis were performed on the full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | HNSCC (IO Naive) | HNSCC (IO Treated) | ESCC | PDAC | Biliary Tract Cancer (BTC) | GBM/AA
Number analyzed (Participants) | 30 | 20 | 30 | 20 | 45 | 30
Participants
  Any AE | 30 | 20 | 30 | 20 | 45 | 30
  Worst grade: Grade 1 | 1 | 0 | 2 | 0 | 1 | 0
  Worst grade: Grade 2 | 4 | 1 | 6 | 2 | 9 | 8
  Worst grade: Grade 3 | 16 | 16 | 18 | 11 | 23 | 11
  Worst grade: Grade 4 | 6 | 2 | 2 | 2 | 1 | 2
  Worst grade: Grade 5 (death) | 3 | 1 | 2 | 5 | 11 | 9

ADVERSE EVENTS:
Time Frame: Up to the last participant has been followed for approximately 10 months, summed up to approximately 26 months
Description: AEs were considered to be treatment-emergent (TEAEs) if they started or worsened after the start of first study drug administration until 30 days after regorafenib treatment discontinuation or 100 days after the last dose of nivolumab, whatever occurred later.
Arm/Group | HNSCC (IO Naive) | HNSCC (IO Treated) | ESCC | PDAC | Biliary Tract Cancer (BTC) | GBM/AA
All-Cause Mortality (participants affected / at risk) | 22/30 | 17/20 | 20/30 | 17/20 | 36/45 | 27/30
Serious Adverse Events (participants affected / at risk) | 22/30 | 15/20 | 19/30 | 13/20 | 28/45 | 13/30
Other Adverse Events (participants affected / at risk) | 30/30 | 20/20 | 30/30 | 20/20 | 45/45 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HNSCC (IO Naive) (N=30) | HNSCC (IO Treated) (N=20) | ESCC (N=30) | PDAC (N=20) | Biliary Tract Cancer (BTC) (N=45) | GBM/AA (N=30)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Oral cavity fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 7 (7) | 9 (10)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (5) | 4 (7) | 4 (6) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 2 (7) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Oral infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Medical device site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crystal arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hemiplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasogenic cerebral oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (5) | 0 (0)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bile duct stent insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Device deposit issue (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HNSCC (IO Naive) (N=30) | HNSCC (IO Treated) (N=20) | ESCC (N=30) | PDAC (N=20) | Biliary Tract Cancer (BTC) (N=45) | GBM/AA (N=30)
Anaemia (Blood and lymphatic system disorders) | 10 (24) | 3 (7) | 5 (12) | 6 (16) | 7 (8) | 2 (3)
Eosinophilia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (4) | 0 (0) | 1 (1) | 3 (6) | 9 (11) | 5 (9)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 5 (6) | 1 (1) | 2 (2) | 1 (1) | 6 (6) | 1 (1)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (6) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (6) | 5 (6) | 8 (10) | 3 (3) | 5 (7) | 3 (3)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 4 (5) | 7 (13) | 11 (16) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 5 (5) | 2 (3) | 8 (12) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Aptyalism (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 7 (8) | 8 (10) | 7 (10) | 7 (9) | 15 (20) | 11 (15)
Diarrhoea (Gastrointestinal disorders) | 7 (10) | 3 (6) | 11 (25) | 3 (5) | 17 (31) | 6 (11)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (5) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 2 (2)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 4 (4) | 2 (2) | 1 (2) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 5 (6) | 7 (10) | 14 (19) | 4 (4)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (7) | 0 (0) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 5 (16) | 3 (7) | 3 (8) | 1 (4) | 3 (4) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 5 (8) | 8 (9) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral cavity fistula (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 10 (17) | 2 (6) | 7 (24) | 4 (6) | 12 (36) | 10 (14)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 2 (2) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (5) | 7 (16) | 9 (19) | 8 (18) | 19 (43) | 5 (10)
Generalised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 4 (9) | 1 (2) | 4 (14) | 1 (1) | 5 (8) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 1 (2) | 2 (2) | 4 (6) | 1 (1)
Pain (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 1 (2)
Pyrexia (General disorders) | 6 (6) | 6 (10) | 12 (20) | 7 (14) | 17 (43) | 5 (6)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 4 (9) | 5 (9)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 1 (2) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 1 (2)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 2 (8) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (3) | 2 (2) | 4 (8) | 0 (0) | 2 (3) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 3 (4) | 1 (1)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acinetobacter bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 4 (4) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 7 (14) | 2 (8) | 4 (10) | 2 (5) | 4 (7) | 3 (12)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 5 (10) | 2 (6) | 3 (6) | 1 (2) | 5 (9) | 4 (12)
Blood bilirubin increased (Investigations) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 6 (10) | 6 (11)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Blood thyroid stimulating hormone increased (Investigations) | 1 (6) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 1 (1) | 3 (6) | 0 (0) | 2 (4) | 6 (13)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (12)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 2 (2) | 3 (5) | 0 (0) | 3 (5) | 3 (4)
Weight decreased (Investigations) | 6 (11) | 3 (3) | 6 (7) | 2 (3) | 5 (6) | 1 (2)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical condition abnormal (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (6) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (2) | 6 (10)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (6) | 0 (0) | 4 (9) | 5 (8) | 5 (10) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2) | 1 (2) | 0 (0) | 4 (4) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (9) | 1 (1) | 4 (4) | 1 (1) | 5 (6) | 1 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 3 (6) | 1 (1) | 4 (8) | 2 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 5 (5) | 1 (1)
Refeeding syndrome (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cell death (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 9 (16) | 11 (26) | 7 (10) | 14 (25) | 6 (10)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Steroid diabetes (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amyotrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 5 (6) | 1 (1) | 6 (8) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 10 (12) | 2 (2)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (2) | 2 (4) | 7 (10) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 5 (8) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 3 (6) | 1 (1)
Sarcopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (10) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Peritumoural oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Apraxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (4)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (5) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Headache (Nervous system disorders) | 1 (2) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 6 (13)
Hemianopia homonymous (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 4 (4) | 2 (2) | 3 (3) | 7 (8) | 3 (3)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (6) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (5) | 4 (4) | 1 (2) | 0 (0) | 0 (0) | 2 (4)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 4 (5) | 2 (3) | 4 (4) | 3 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 5 (6) | 3 (3) | 9 (9) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (7) | 2 (2) | 5 (7) | 1 (1) | 4 (6) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 5 (10) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 6 (6) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 8 (11) | 9 (28) | 22 (45) | 5 (16) | 15 (37) | 8 (18)
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3) | 3 (4) | 1 (2) | 5 (5) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 6 (7) | 2 (2) | 14 (23) | 8 (14) | 10 (22) | 5 (8)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 5 (8) | 1 (2)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Scar pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 5 (7) | 7 (12) | 4 (7) | 6 (13) | 11 (25) | 8 (16)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/54/NCT04704154/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT04704154/SAP_002.pdf